CLINICAL TRIAL: NCT00665496
Title: A Randomized, Double Blind, Double Dummy, Parallel Group, Multi-center Study to Investigate the Time to Onset of Action of 10 mg and 20 mg of Vardenafil Compared to Placebo in Males With Erectile Dysfunction.
Brief Title: A Study to Investigate the Time to Onset of Action of 10 mg and 20 mg of Vardenafil Compared to Placebo in Males With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100492; ONTIME
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil; Onset of action
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 10 mg and 20 mg orally once a day as needed
  Arms: Arm 1
Drug: Placebo — Matching Placebo
  Arms: Arm 2

SUMMARY:
This purpose of the study was to evaluate the earliest time to onset of action in adults with erectile dysfunction (often called impotence). In this study vardenafil has been compared to placebo. Patients were asked to fill in questionnaires and a diary in which they filled in details about attempts at sexual activity during study period. Patients received also a stopwatch to record the time of onset of erection. Stopwatch should be started immediately prior to initiating sexual activity and stopped when an erection perceived to be adequate for penetration was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Males with ED for more than 6 months according to the NIH Consensus statement(inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance)
* Heterosexual relationship
* 18 years and older

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life threatening arrhythmia within the prior 6 months
* Nitrates or nitric oxide donors use
* Other exclusion criteria according to the US Product Information

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2003-06; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
- Earliest elapsed time from dosing to attainment of an erection perceived to be adequate for penetration leading to completion of successful intercourse as measured by Sexual Encounter Profile Question 3 (SEP 3) | First four doses with successful intercourse

SECONDARY OUTCOMES:
- Earliest elapsed time from dosing to attainment of an erection perceived to be adequate for penetration as measured by Sexual Encounter Profile Question 2 (SEP 2). | among the first four doses
- The erectile function (EF) domain score of the International Index of Erectile Function (IIEF) calculated as the sum of scores from Questions 1-5 and 15 at Week 4 as well as all other IIEF factor subscores. | among the first four doses
- Responder time to onset, where onset is time from dosing to attainment of an erection perceived to be adequate for penetration. | among the first four doses
- Other diary questions | among the first four doses
- Safety and tolerability | within the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (71):
- United States (12):
  - Phoenix, Arizona
  - Beverly Hills, California
  - San Bernardino, California
  - Aurora, Colorado
  - Trumbull, Connecticut
  - Aventura, Florida
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - Lawrenceville, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Wilmington, North Carolina
- Canada (8):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - Kentville, Nova Scotia
  - Barrie, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- France (7):
  - Carpentras
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nîmes
  - Paris
- Germany (12):
  - Garmisch-Partenkirchen, Bavaria
  - München, Bavaria
  - Hamburg, Hamburg
  - Marburg, Hesse
  - Hanover, Lower Saxony
  - Osnabrück, Lower Saxony
  - Westerstede, Lower Saxony
  - Düsseldorf, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Niederkassel, North Rhine-Westphalia
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
- Italy (4):
  - Milan
  - Modena
  - Napoli
  - Padua
- Netherlands (5):
  - Amsterdam
  - Nijmegen
  - Roermond
  - The Hague
  - Utrecht
- Norway (4):
  - Moelv
  - Oslo
  - Sarpsborg
  - Trondheim
- Poland (6):
  - Warsaw, Poland
  - Kościerzyna
  - Lodz
  - Poznan
  - Warsaw
  - Wroclaw
- Spain (8):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Galdakao, Bizkaia
  - Castellon, Castellón de La Plana
  - Barcelona, Catalonia
  - Madrid, Madrid
  - Zaragoza, Zaragoza
- Sweden (4):
  - Borås
  - Gothenburg
  - Skövde
  - Stockholm
- Bristol, Avon, United Kingdom